CLINICAL TRIAL: NCT02343601
Title: Perioperative Hemodynamic Optimization Using the Photoplethysmography in Colorectal Surgery : A Randomized Controlled Study
Brief Title: Perioperative Hemodynamic Optimization Using the Photoplethysmography in Colorectal Surgery
Acronym: PANEX3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2014-A00870-47
Record Dates: First submitted 2014-06-13; First posted 2015-01-22 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Polyp of Large Intestine; Colorectal Neoplasms; Crohn Disease
MeSH Terms: conditions — Colorectal Neoplasms; Crohn Disease | interventions — Photoplethysmography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control group using a hemodynamic standard protocol
- Photoplethysmography group (Other): Hemodynamic optimization using Photoplethysmography device (ClearSight, Edwards Lifesciences, Irvine, CA)
  Interventions: Device: Photoplethysmography

INTERVENTIONS:
Device: Photoplethysmography — Use Photoplethysmography for hemodynamic optimization during colorectal perioperative period
  Arms: Photoplethysmography group

SUMMARY:
The purpose of this study is to determine whether hemodynamic optimization with photoplethysmography (ClearSight, Edwards Lifesciences, Irvine, CA) during colorectal surgery could decrease the incidence of perioperative complications.

DETAILED DESCRIPTION:
All patients received the photoplethysmography monitoring, but the monitor was blinded in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Colorectal surgery

Exclusion Criteria:

* Pregnant women
* Black skin
* Chronic renal insufficiency (MDRD <30 ml/min)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of patients presenting at least one complication after colorectal surgery | Up to 28 days after surgery (length of hospital stay)
  Two independent experts defined the presence of complication using an a priori classification.

SECONDARY OUTCOMES:
All complications happening after colorectal surgery | Up to 28 days after surgery (length of hospital stay)
Real length of hospital stay | Up to 28 days after surgery (length of hospital stay)
Perioperative mortality | 28 days after surgery

OTHER OUTCOMES:
Medico economic evaluation of cost of treatment | Up to 28 days after surgery (length of hospital stay)
  Medico economic evaluation of photoplethysmography use will be assessed with a specific unit of measure, using cost of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Fiant, MD, Principal Investigator — University Hospital of Caen
Locations (1):
- Caen University Hospital, Caen, France

REFERENCES:
- [Derived] Fischer MO, Fiant AL, Boutros M, Flais F, Filipov T, Debroczi S, Pasqualini L, Rhanem T, Gerard JL, Guittet L, Hanouz JL, Alves A, Parienti JJ; PANEX3 study group. Perioperative hemodynamic optimization using the photoplethysmography in colorectal surgery (the PANEX3 trial): study protocol for a randomized controlled trial. Trials. 2016 Mar 22;17:159. doi: 10.1186/s13063-016-1278-4. PMID 27004412